CLINICAL TRIAL: NCT06660277
Title: DIALysis With EXpanded Solute Removal (DIALEX): A Large, Simple Randomized Trial to Evaluate the Major Health Effects of Expanded Versus Conventional Hemodialysis.
Brief Title: DIALysis With EXpanded Solute Removal
Acronym: DIALEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Schulich School of Medicine and Dentistry (Unknown); ICES (Industry); Nipro Canada Corporation (Unknown); London Health Sciences Centre (Other); Statistics Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4954; R-25-209 (Other: London Health Sciences Centre)
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis; End-Stage Kidney Disease (ESKD); Chronic Kidney Disease Requiring Chronic Dialysis; Pragmatic Randomized Controlled Trial; Kidney Disease; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Hemodialysis
Keywords: Nipro Elisio HX; RCT; Dialyzer; Hemodialysis Filter; Super-High Flux Dialyzer; High-Flux Dialyzer; Expanded Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:3 or 1:1 (Expanded HD : Conventional High-Flux HD) ratio, depending on their study site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expanded Hemodialysis (Experimental): Participants will receive their regularly scheduled hemodialysis treatments using a super high-flux dialyzer (Nipro Elisio HX).
  Interventions: Device: Super High-Flux Dialyzer
- Conventional Hemodialysis (Active Comparator): Participants will receive their regularly scheduled hemodialysis treatments using a high-flux dialyzer (as prescribed in routine care).
  Interventions: Device: High-Flux Dialyzer

INTERVENTIONS:
Device: Super High-Flux Dialyzer — A hemodialysis filter (known as a dialyzer) that is currently approved by Health Canada and available for use across Canada. This filter has larger pores than a high-flux dialyzer that allow for greater removal of potential toxins and wastes in the blood that would regularly be filtered out by healthy kidneys.
  Other Names: Expanded Hemodialysis; Nipro Elisio HX; Sharp Cut-Off Dialyzer; Medium Cut-Off Dialyzer
  Arms: Expanded Hemodialysis
Device: High-Flux Dialyzer — A hemodialysis filter (known as a dialyzer) that is that is widely used across Canada for hemodialysis treatments.
  Other Names: Conventional Hemodialysis
  Arms: Conventional Hemodialysis

SUMMARY:
The goal of this clinical trial is to evaluate the health effects of expanded hemodialysis in patients receiving hemodialysis. The main question it aims to answer is:

1) Does expanded hemodialysis reduce the risk of death from any cause?

Researchers will compare expanded hemodialysis to conventional hemodialysis (the treatment currently used for the majority of patients receiving hemodialysis) to see if expanded hemodialysis works to improve patient outcomes.

Participants will continue to receive their regularly scheduled hemodialysis treatments using either a super high-flux/expanded dialysis filter or a high-flux/conventional dialysis filter. All other aspects of treatments remain the same. No additional tests or visits are required. Data will be obtained using administrative healthcare databases and medical record review (at a subset of participating locations).

DETAILED DESCRIPTION:
Background:

Expanded hemodialysis refers to hemodialysis treatment using a newer generation of hemodialysis filters or "dialyzers" that remove large middle molecules to a greater extent than conventional "high-flux" dialyzers. This is expected to improve major health outcomes. However, despite a decade of availability and promising surrogate data from small trials and patient outcomes data from large observational studies, dialyzers capable of providing expanded hemodialysis have failed to achieve significant adoption conventional high-flux dialyzers in the absence of more definitive evidence. A large, rigorous randomized controlled trial is necessary to establish the clinical effectiveness of expanded hemodialysis compared to conventional hemodialysis with high-flux dialyzers.

Study Design:

Parallel, block randomized, controlled, open label, superiority trial comparing the clinical effects of expanded hemodialysis using Nipro Elisio HX dialyzers to conventional hemodialysis using high-flux dialyzers. The allocation ratio will vary between 1:3 or 1:1 ratio depending on their dialysis unit.

Setting:

Community and academic hemodialysis facilities.

Study Size:

4800 participants (1200 in expanded hemodialysis arm and 3600 in conventional high-flux hemodialysis arm) followed for a mean of 2.9 years.

Trial Duration:

Duration of participant accrual - 2 years from date of first participant recruited.

Total duration - 5 years from date of first participant recruited. Trial results anticipated to be announced in 2030.

Study Power:

90% power to detect 15% relative reduction in the hazard of death (hazard ratio 0.85).

ELIGIBILITY:
Inclusion Criteria: Inclusion requires that all the following are present:

1. One of:

   1. Age 60 years or older; or
   2. Age 45 to 59 years with a history of diabetes mellitus (Type 1 or Type 2) regardless of current glycemic status; and
2. Receiving any form of dialysis regularly for the previous 90 days; and
3. Currently receiving HD in-centre (main or satellite unit) 3 or more times per week; and
4. A valid provincial or territorial health insurance card number.

Exclusion Criteria: Patients are ineligible if they meet any of the following criteria:

1. Not appropriate for this study in the opinion of the treating nephrologist or dialysis nurse practitioner due to any of:

   1. Known or anticipated intolerance to the Nipro Elisio HX dialyzer; or
   2. Planned to receive HDF; or
   3. Planned to receive nocturnal HD; or
   4. Anticipated to discontinue in-centre HD in the next 3 months for any reason (examples: palliation, transplantation, home dialysis, recovery of kidney function, death, others); or
   5. Anticipated severe non-adherence to the frequency or duration of prescribed dialysis treatment; or
   6. An overriding clinical preference for expanded HD (i.e., dialysis with the Elisio HX or other comparable dialyzer, such as Baxter TheranovaTM); or
   7. Another medical, psychosocial, or logistical reason; or
2. Enrolled in another clinical trial that explicitly prohibits concurrent participation in other clinical trials or that would substantially interfere with adherence to the DIALEX procedures (note that DIALEX otherwise permits concurrent participation in other trials); or
3. Previously enrolled in this trial; or
4. Declined participation.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome of All-Cause Mortality | From randomization to event (death) or end of treatment (average 2.9 years follow-up), whichever occurs first
  Outcome data will be collected as a result of routine patient interactions with the healthcare system and will be obtained from national and provincial data repositories (with the exceptions of routine care symptoms and ESA utilization outcomes, in participating sites), enabling health records to be analyzed in a privacy-compliant manner. These datasets have high levels of completeness and validity. The primary outcome, all-cause mortality, is captured with over 99% accuracy in our data sources.

SECONDARY OUTCOMES:
Key Secondary Outcome of Cardiovascular and Infection-Related Hospitalizations | From randomization to the end of treatment (average 2.9 year follow-up)
  The key secondary outcome will be time to first and recurrent cardiovascular or infection-related hospitalizations. Cardiovascular and infection-related hospitalizations will be ascertained using primary discharge ICD-10 diagnosis codes in the Canadian Institute for Health Information Discharge Abstract Database
Cardiovascular-Related Hospitalizations | From randomization to the end of treatment (average 2.9 year follow-up)
  Time to first and recurrent cardiovascular hospitalizations. Each component of the secondary outcome (cardiovascular-related and infection-related hospitalizations) will be examined separately.
Infection-Related Hospitalizations | From randomization to the end of treatment (average 2.9 year follow-up)
  Time to first and recurrent infection-related hospitalizations. Each component of the secondary outcome (cardiovascular-related and infection-related hospitalizations) will be examined separately.
Death from Cardiovascular Cause | From randomization to end of treatment (average 2.9 year follow-up).
  Defined as any out-of-hospital death or death that occurred during a hospitalization for a cardiovascular cause captured in Canada in the CIHI-DAD database.
Death from Non-cardiovascular Cause | From randomization to end of treatment (average 2.9 year follow-up).
  Death that does not meet the definition for death from a cardiovascular cause.
Receipt of a Functional Kidney Transplant | From randomization to event (functioning kidney transplant) or end of treatment (average 2.9 years follow-up), whichever comes first.
  Receipt of a functional kidney transplant is defined, in Canada, by a record of a hospital admission in the CIHI-DAD database with an ICD-10 code for kidney transplantation followed by discontinuation of dialysis in the absence of death. Receipt of a functioning kidney transplant refers to the first functioning transplant received after randomization.

OTHER OUTCOMES:
Routine Care Symptoms | From randomization to the end of treatment (average 2.9 year follow-up)
  Routine care symptoms assessed using the Edmonton Symptoms Assessment System Revised Renal (ESAS-r: Renal) instrument, as recorded in usual care. Data will be abstracted from routine clinical records. The ESAS-r: Renal evaluates 12 symptoms on a 0-10 scale, with assessments every 3-6 months. The minimum value is 0, meaning no experience of specified symptom. The maximum value is 10 meaning, worst possible experience of specified symptom. This will be done only in units that routinely administer this instrument and participation in reporting this outcome is optional for sites.
Healthcare-Associated Costs | From randomization to the end of treatment (average 2.9 year follow-up)
  The investigator will assess healthcare-associated costs in the subset of patients enrolled in Ontario using linked administrative databases with a standard method developed by the Institute for Clinical Evaluative Sciences (ICES).
Neutrophil to Lymphocyte Ratio | From randomization to the end of treatment (average 2.9 year follow-up)
  The ratio between the neutrophil count and lymphocyte count derived from a complete blood count measurement performed in routine care and captured in the Ontario Laboratory Information System. This measures is typically collected every 4-6 weeks as part of standard dialysis care in Ontario.
Blood Hemoglobin Concentration | From randomization to end of treatment (average 2.9 years follow-up)
  Hemoglobin concentration from a complete blood count measurement performed in routine care and captured in the Ontario Laboratory Information System. This measures is typically collected every 4-6 weeks as part of standard dialysis care in Ontario.
Serum Albumin Concentration | From randomization to the end of treatment (average 2.9 year follow-up)
  Serum albumin concentration measured in routine care and captured in the Ontario Laboratory Information System. This measures is typically collected every 4-6 weeks as part of standard dialysis care in Ontario.
Erythropoietin Stimulating Agent (ESA) Utilization | From randomization to end of treatment (average 2.9 years follow-up)
  ESAs include darbepoetin or epoetin. Doses will be expressed as the dose per week. Dose will be converted to the weekly total epoetin dose and expressed as units per week. Subcutaneous and intravenous dosing will be considered equivalent. Data will be obtained from local medical record review and reported approximately every 6 months. Participation in reporting of this outcome is optional for sites and will only be assessed in a subset of participating sites.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel S Roshanov, MD MSc FRCPC, Principal Investigator — London Health Sciences Centre Research Institute; Amit X Garg, MD PhD FRCPC FACP, Study Chair — London Health Sciences Centre Research Institute
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No